CLINICAL TRIAL: NCT02589561
Title: REFIT Hearing: Remote Fitting of Hearing Aids
Acronym: REFITHEARING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: AudioPro Connect (Industry); Alliance Audition Montpellier (Other); Audition Conseil Perpignan (Other); Audition Conseil à Nîmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 9594
Record Dates: First submitted 2015-10-21; First posted 2015-10-28 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Hearing Loss
Keywords: hearing loss; hearing aids
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- face to face fitting (Active Comparator): face to face fitting of hearing aids
  Interventions: Device: Remote fitting; Device: Face to face fitting
- remote fitting (Experimental): remote fitting of hearing aids
  Interventions: Device: Remote fitting; Device: Face to face fitting

INTERVENTIONS:
Device: Remote fitting — remote fitting of hearing aids
Device: Face to face fitting — face to face fitting of hearing aids

SUMMARY:
Currently, the fitting of hearing aids is using a computer interface that allows to adjust the gain and compression of acoustic amplification. This adjustment is made face to face, patient and audiologist being located in a soundproof space to test the effectiveness of the hearing aid.

However, advances in telemedicine in this context, let consider the possibility of addressing these hearing aids fitting via the same computer interface, but remotely controlled by the hearing care professional. The purpose of this study is to assess the ability to perform these tests no longer in front of the patient settings, but away from it, and without visual and sound contact other than through a computer interface.

At the end, this project wants to show that a remote fitting is an acceptable procedure that provides comparable results to-face fitting in terms of speech perception, speech in noise audiometry, hearing loss related quality of life in order to be able to offer this type of strategy.

DETAILED DESCRIPTION:
1. Background and rationale:

   Currently, the fitting of hearing aids is using a computer interface that allows to adjust the gain and compression of acoustic amplification. This adjustment is made face to face, patient and audiologist being located in a soundproof space to test the effectiveness of the hearing aid.

   However, advances in telemedicine in this context, let consider the possibility of addressing these hearing aids fitting via the same computer interface, but remotely controlled by the hearing care professional. The purpose of this study is to assess the ability to perform these tests no longer in front of the patient settings, but away from it, and without visual and sound contact other than through a computer interface.
2. Objectives Main objective: To show that the remote fitting of hearing aids using the platform developed by AudioProConnect provides speech perception scores similar to those obtained by a face-control, after 5 weeks of use among experienced hearing aid users.

   Secondary Objectives: To compare the duration and the quality of both types of fitting, speech in noise testing, deafness related quality of life and assess the wearing time of hearing aids.
3. Methods DESIGN: Biomedical research on health product, prospective, multicenter, randomized, and crossover study to assess the remote fitting of hearing aids: Study REFIT-HEARING Study Population: adults with bilateral hearing aids. Inclusion criteria: Patient aged between 18 and 85 years old, with hearing loss and using two hearing aids for more than one year, and compatible with AudioProConnect platform.

   Exclusion criteria: Patient with fluctuations of pure tone audiometry, cognitive disorders or severe speech disorders. Patient unable to move in an audiology laboratory.

   Primary Outcome: Evaluation of speech perception score with PBK test free-field at 60 dB.

   Secondary endpoints: assessment of quality control by measuring the pitch gain, duration of fitting in minutes, speech in noise audiometry, the wearing time of hearing aids in hours, the quality of life related to hearing loss via the APHAB questionnaire.

   Number of patients: 60 subjects Procedure (number of visits, length of inclusions, duration of follow-up, study schedule patient visits content, brief description of intervention): After the investigator has verified the criteria of inclusion / non inclusion and the subject has signed the written informed consent, the subject will be followed for a period ranging from 2 months to 5 months, during which he attended four visits in a audiology laboratory referenced in this project. During these visits, a fitting of hearing aids face to face or remotely will be realized, and it will be asked to answer a questionnaire to assess quality of life between the two fitting techniques.

   Study Schedule:

   Inclusion period: 3 months (M3-M6) Duration of the study for one subject: 2 months to 5 months (M6 to M8 or M6 to M11) Duration statistical analysis / recovery: 3 months (M11-M14) Global Study duration: 14 months
4. Outlook At the end, this project wants to show that a remote fitting provides comparable results to-face fitting in terms of speech perception, in order to be able to offer this type of strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age limits ≥ 18 et < 85 years
* User of two hearing aids for more than a year
* Carriers of adjustable digital hearing aids by means of a software of the usable manufacturer on Windows® PC (in stand-alone or as plug-in in the software NOAH®) to be integrated into the platform AudioProConnect. It is the case of almost all the current hearing aids (Phonak, Starkey, Siemens, Unitron, etc.)
* Subject able to understand the nature, the aim and the methodology of the study.
* Affiliation or recipient with the mode of social security.
* Collection of the informed consent

Exclusion Criteria:

* Fluctuations in the tonal audiometry, defined as variations furthermore of 10 dB of the average hearing loss (Average arithmetic of thresholds in 500, 1000, 2000 et 4000 Hz) Between the last 2 tonal audiometries realized over the previous 2 years
* Cognitive disorders or severe phasic hampering the understanding of the language or the repetition of the speech (Subject not being capable of participating in a vocal audiometry during the last regulation of its hearing aids)
* Incapacitated to move in a laboratory of audioprosthesis
* Fickle bearing of the hearing aid (<6h /day ou < 5day/7)
* Tip not adapted little finger
* Presence of plugs of earwax at the time of the tests
* Patient minor(miner) or protected adults or in the incapacity to give its consent according to the article L1121-8 Of the Public Code of the Health (CSP)
* Pregnant or breast-feeding women according to the article L1121-5 du CSP.
* Vulnerable people according to the article L1121-6 du CSP.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
speech perception | 5 months
  score PBK test

SECONDARY OUTCOMES:
speech in noise audiometry | 5 months
quality of life | 5 months
  APHAB questionnaire
duration of fitting | 5 months
daily use of hearing aids | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric VENAIL, Professor, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Hôpital Gui de Chauliac - Service ORL, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Venail F, Picot MC, Marin G, Falinower S, Samson J, Cizeron G, Balcon M, Blanc D, Bricaud J, Lorenzi A, Ceccato JC, Puel JL. Speech perception, real-ear measurements and self-perceived hearing impairment after remote and face-to-face programming of hearing aids: A randomized single-blind agreement study. J Telemed Telecare. 2021 Aug;27(7):409-423. doi: 10.1177/1357633X19883543. Epub 2019 Nov 6. PMID 31694484